CLINICAL TRIAL: NCT05573971
Title: The Effect of Verbal Encouragement on Performance and Muscle Fatigue in Swimming
Brief Title: Verbal Encouragement in Swimming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Luca Puce, Principal Investigator, Universita degli Studi di Genova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VES-DINOGMI-21
Record Dates: First submitted 2022-09-30; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: verbal encouragement; performance; muscle fatigue; swimming; sEMG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with verbal encouragement (Experimental)
  Interventions: Other: with verbal encouragement
- without verbal encouragement (No Intervention)

INTERVENTIONS:
Other: with verbal encouragement — Each athlete swam a maximal 200m freestyle trial in two different conditions: one trial with verbal encouragement and the other without verbal encouragement
  Arms: with verbal encouragement

SUMMARY:
Verbal encouragement (VE) is used to enhance the performance in several sports, even though no studies have been conducted in swimmers and no effects have been reported in elite athletes by some Authors. Besides influencing motor performance, VE is also known to enhance the physical load, thus increasing the probability of developing fatigue. The aim of this research was to study VE in swimmers by evaluating both chronometric performance and muscle fatigue (using sEMG).

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year of experience in training aimed at regional and international competitions
* a score ≥ 200 points on the personal best in the 200m freestyle, in accordance with the international point score (IPS) (http://www. swimnews.com/ipspoints)
* being healthy

Exclusion Criteria:

* having a disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
swimming velocity | up to 2min 30s
  m/sec

SECONDARY OUTCOMES:
Pectoralis Major muscle fatigue | up to 2min 30s
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal measured for Pectoralis Major muscle
Triceps Brachii muscle fatigue | up to 2min 30s
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal measured for Triceps Brachii muscle
Latissimus Dorsi muscle fatigue | up to 2min 30s
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal measured for Latissimus Dorsi muscle
Rectus Femoris muscle fatigue | up to 2min 30s
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal measured for Rectus Femoris muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Genova, Genoa, GE, Italy

IPD SHARING:
Plan to Share IPD: No